CLINICAL TRIAL: NCT05690009
Title: Real Clinical Practice Register of AlbUminuRia Detection in Patients With Previously undiAgnosed Chronic Kidney Disease
Acronym: AURA
Status: Completed | Type: Observational
Sponsor: Eurasian Association of Therapists (Other)
Responsible Party: Sponsor
Other Study IDs: AURA
Record Dates: First submitted 2022-12-29; First posted 2023-01-19 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Hypertension; Chronic Heart Failure; Ischemic Heart Disease; Atrial Fibrillation; PreDiabetes; Chronic Obstructive Pulmonary Disease; Cancer; Urolithiasis; COVID-19
Keywords: Albumin-to-creatinine ratio; Albuminuria; Microalbuminuria; Chronic Kidney Diseases; Estimation of glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Myocardial Ischemia; Atrial Fibrillation; Prediabetic State; Pulmonary Disease, Chronic Obstructive; Neoplasms; Urolithiasis; COVID-19; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with albuminuria: Patients aged 40 or older without preexisting diagnoses of chronic kidney disease, type 1 diabetes, and type 2 diabetes with positive albuminuria by dipsticks and/or microalbuminuria test or albumin-to-creatinine ratio in a single urine sample.

SUMMARY:
Real clinical practice register of Albuminuria detection in patients with previously undiagnosed chronic kidney disease

DETAILED DESCRIPTION:
This register was sponsored and organized by the Association "Eurasian Association of Internal Medicine". It is a multicenter non-interventional register of real clinical practice. The database will include patients aged 40 years and older without pre-existing nephrological disease who are available for a dipstick test for albuminuria. The subjects will be identified by screening all patients who meet inclusion/exclusion criteria during routine outpatient and hospital follow-up. The register does not include follow-up (cross-sectional design).

Patients eligible for the register should be enrolled and documented. The procedure for obtaining informed consent for the collection and analysis of the retrospective data must comply with the local legislation. If necessary, patients will be asked to sign an informed consent document.

All study sites will use standardized electronic CRFs. The Electronic Data Capture (EDC) system should be validated in accordance with current standards and legal requirements. The investigators will log into this system using individual usernames and passwords. Data may only be entered and corrected by the investigator or other authorized study site personnel.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 and older at the time of data entry;
* A possibility to check for albuminuria using dipsticks and/or analysis for microalbuminuria or albumin-to-creatinine ratio in a single urine sample.

Exclusion Criteria:

* Unwillingness of the patient to participate in the register;
* Diagnosis of CKD made before the screening for the register;
* Diagnosis of diabetes mellitus (DM) type 1 or type 2 made before the screening for the register;
* Pregnancy;
* Long distance running or very strenuous physical activity in the last 24 hours.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 40 or older without preexisting diagnoses of chronic kidney disease, type 1 diabetes, and type 2 diabetes will be enrolled into this register.
Sampling Method: Probability Sample
Enrollment: 4580 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of AU and its severity. | Day 1
  Determination of AU by qualitative and/or quantitative methods

SECONDARY OUTCOMES:
Number of comorbidities per patient with AU. | Day 1
  Number of comorbidities per patient with AU.
Frequency of prescribing renoprotective drugs. | Day 1
  Frequency of prescribing renoprotective drugs.
Calculation of eGFR according to CKD-EPI formula 2021 in different phenotypes from the study population. | Day 1
  Calculation of eGFR according to CKD-EPI formula 2021 in different phenotypes from the study population.
Prevalence of probable CKD in the study sample based on the clinical and laboratory data obtained during the screening. | Day 1
  Prevalence of probable CKD in the study sample based on the clinical and laboratory data obtained during the screening.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Arutyunov, professor, Study Chair — Eurasian Association of Internal Medicine
Locations (1):
- Eurasian Association of Therapists, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No